CLINICAL TRIAL: NCT05373953
Title: Open-label, Non-randomised, Parallel-group Study to Investigate the Pharmacokinetics, Safety and Tolerability Following Single Administration of CHF6001 in Subjects With Mild, Moderate and Severe Liver Impairment in Comparison With Matched Healthy Control Subjects
Brief Title: Clinical Study to Investigate the Pharmacokinetics, Safety and Tolerability Following Single Administration of CHF6001 in Subjects With Mild, Moderate and Severe Liver Impairment in Comparison With Matched Healthy Control Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CLI-06001AA1-08; 2021-003729-31 (EudraCT Number)
Record Dates: First submitted 2022-05-10; First posted 2022-05-13 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tanimilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- mild impairment subjects (Experimental): Administration of a single dose of CHF6001 800 µg in mild impairment subjects
  Interventions: Drug: CHF6001
- moderate impairment subjects (Experimental): Administration of a single dose of CHF6001 800 µg in moderate impairment subjects
  Interventions: Drug: CHF6001
- severe impairment subjects (Experimental): Administration of a single dose of CHF6001 800 µg in severe impairment subjects
  Interventions: Drug: CHF6001
- healthy volunteers (Active Comparator): Administration of a single dose of CHF6001 800 µg in healthy volunteers
  Interventions: Drug: CHF6001

INTERVENTIONS:
Drug: CHF6001 — CHF6001 will be administered using the NEXThaler® DPI device

SUMMARY:
A clinical trial to investigate the pharmacokinetics, safety and tolerability of CHF6001 after single administrations in participants with mild, moderate and severe liver impairment with matched healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

* All subjects:

  1. Subject's written informed consent obtained prior to any study-related procedure;
  2. Ability to understand the study procedures and the risks involved, and ability to be rained to use the inhalers correctly and to generate sufficient peak inspiratory flow (PIF; at least 40 L/min) using the In- Check DIAL set as per NEXThaler® inhaler resistance;
  3. 12-Lead digitised electrocardiogram (ECG) in triplicate considered as normal (40 beats per minute [bpm] ≤ heart rate [HR] ≤ 110 bpm, 120 ms ≤ PR interval [PR] ≤ 210 ms, QRS interval [QRS] ≤ 120 ms, QT Interval corrected using Fridericia's formula [QTcF] ≤ 450 ms for males and QTcF ≤ 470 ms for females) at screening visit. The mean value must be within the defined range;
  4. Male and female subjects aged 40 to 80 years inclusive;
  5. Subjects must weigh at least 45 kg for females and 50 kg for males to participate in the study, and must have a body mass index within the range of 18 to 35 kg/m2 inclusive;
  6. Non- or ex-smokers who smoked < 5 pack-years (pack-years = the number of cigarette packs per day times the number of years) and stopped smoking > 1 year prior to screening;
  7. Female subjects: a. Women of childbearing potential (WOCBP) fulfilling one of the following criteria: i. WOCBP with fertile male partners: they and/or their partner must be willing to use at least an acceptable effective birth control method from the signature of the informed consent and until study discontinuation; or ii. WOCBP with non-fertile male partners (contraception is not required in this case); b. Female subjects of non-childbearing potential defined as physiologically incapable of becoming pregnant (i.e. post-menopausal or permanently sterile. Tubal ligation or partial surgical interventions are not acceptable.
  8. Vital signs within normal limits at screening: diastolic blood pressure (DBP) 40-89 mmHg and systolic blood pressure (SBP) 90-139 mmHg, extremes included (two measures performed after at least 5 minutes of resting).
  9. Body temperature < 37.5°C at screening and prior to study treatment administration;
  10. Lung function measurements within normal limits at screening: forced expiratory volume within the first second (FEV1) > 80% predicted and FEV1/forced vital capacity (FVC) ratio > 0.70;

      Healthy subjects only:
  11. Good mental and physical status, determined on the basis of the medical history and a general clinical examination, at screening and prior to study treatment administration;
  12. Matched to at least one liver impaired subject enrolled in the study with respect to race, gender, age (±10 years) and body weight (±15%)

      Liver impaired subjects only:
  13. Documented chronic stable liver disease based on the Child-Pugh score and classification (Child-Pugh Class A [mild], B [moderate] or C [severe]) at screening and on Day -1:
  14. Liver impairment must be caused by hepatic primary disease, not a complication of other underlying diseases.

Exclusion Criteria:

* All subjects:

  1. For females only: pregnant or lactating women, where pregnancy is defined as the state of a female after conception and until termination of the gestation, confirmed by a positive serum human chorionic gonadotropin laboratory test. Serum pregnancy test to be performed at screening and urine pregnancy test to be performed prior to study treatment administration;
  2. Subjects with history of breathing problems (i.e. history of asthma including childhood asthma);
  3. Positive human immunodeficiency virus (HIV) 1 or HIV2 serology at screening;
  4. Subject has pre-planned surgery or procedures that would interfere with the conduct of the study;
  5. Documented coronavirus disease 2019 (COVID-19) diagnosis within the last 8 weeks, or complications from this disease, which has not resolved within 14 days prior to screening or prior to study treatment administration;
  6. Blood donation or blood loss (≥ 450 mL) less than 2 months prior to screening or prior to study treatment administration;
  7. Abnormal haemoglobin level defined as < 13 g/dL for males and < 11 g/dL for females at screening;
  8. Documented history of drug abuse within 12 months prior to screening or a positive urine drug screen evaluated at screening or prior to study treatment administration;
  9. Intake of non-permitted concomitant medications in the predefined period prior to screening or prior to study treatment administration, or the subject is expected to take non-permitted concomitant medications during the study
  10. Unsuitable veins for repeated venepuncture;
  11. Participation in another clinical study where an investigational treatment was received, and last investigations were performed less than 8 weeks prior to screening;
  12. Presence of any current infection, or previous infection that resolved less than 7 days prior to screening or to study treatment administration;
  13. Known intolerance and/or hypersensitivity to any of the excipients contained in the formulation used in the study;
  14. Heavy caffeine drinker (average of > 5 cups or glasses per day of caffeinated beverages e.g. coffee, tea, cola, calculated by number of standard espresso portions);
  15. Positive urine test for cotinine at screening or prior to study treatment administration;
  16. Contra-indications/warnings/precaution for use: contra-indications to the investigational medicinal product constitute an exclusion criterion. For warnings/precaution for use, eligibility will be judged by the Investigator;
  17. The use of any kind of smoking electronic devices within 6 months before screening and before study treatment administration;
  18. Clinically relevant and/or uncontrolled cardiovascular, renal, gastrointestinal, haematological, endocrine, metabolic, respiratory, neurologic, neoplastic or psychiatric disorder that, based on the Investigator's judgment, may interfere with successful completion of this study.

      Healthy subjects only:
  19. Any hepatic disorder that, based on the Investigator's medical judgment, may interfere with successful completion of this study;
  20. Positive results from the hepatitis serology which indicate acute or chronic hepatitis B or hepatitis C (e.g. positive hepatitis B surface antigen [HBsAg], hepatitis B core antibody [immunoglobulin M antibody to hepatitis B core antigen; IgM anti-HBc], hepatitis C virus [HCV] antibody); Note: Subjects with an isolated antibody to HBsAg (anti-HBs) positive result, immune due to a medical history of vaccination, are permitted;
  21. Abnormal liver enzymes at screening or prior to study treatment administration (alanine aminotransferase [ALT], aspartate aminotransferase [AST], gamma-glutamyl transpeptidase, alkaline phosphatase or total bilirubin; ALT or AST > 1.5 times the upper limit of normal [ULN], bilirubin > 1.5 times the ULN);
  22. Documented history of alcohol abuse within 12 months prior to screening or a positive alcohol breath test at screening or prior to study treatment administration;
  23. Clinically relevant abnormal laboratory values at screening suggesting an unknown disease and requiring further clinical investigation or which may impact the safety of the subject or the evaluation of the result of the study according to the Investigator's judgment;

      Liver impaired subjects only:
  24. Impaired renal function (estimated glomerular filtration rate [eGFR] < 60 mL/min/1.73 m2) due to primary or secondary renal disease (e.g. hepatorenal syndrome);
  25. Documented history of alcohol abuse within at least 3 months prior to screening or a positive alcohol breath test at screening or prior to study treatment administration;
  26. Severe complications of liver disease within the preceding 3 months prior to enrolment (e.g. Grade 3-4 encephalopathy, severe ascites, severe haemostatic impairment, gastrointestinal haemorrhage, spontaneous bacterial peritonitis or emergency room visit/hospitalisation due to liver disease);

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter (Cmax) | Over 240 hours after administration in blood
  Peak Plasma Concentration (Cmax) for CHF6001 for total plasma
Pharmacokinetic parameter (AUCt) | Over 240 hours after administration in blood
  Area under the plasma concentration versus time curve (AUCt) for CHF6001 for total plasma

SECONDARY OUTCOMES:
Pharmacokinetic parameter ( Cmax) | Over 240 hours after administration in blood
  Peak Plasma Concentration (Cmax) for CHF6001 unbound plasma
Pharmacokinetic parameter (AUCt) | Over 240 hours after administration in blood
  Area under the plasma concentration versus time curve (AUCt) for CHF6001 unbound plasma
Pharmacokinetic parameter (AUC0-72) | Over 72 hours after administration in blood
  Area under plasma concentration from 0 to 72hours (AUC0-72) for CHF6001, CHF5956 and CHF6095
Pharmacokinetic parameter (AUC0-240) | Over 240 hours after administration in blood
  Area under plasma concentration from 0 to 240hours (AUC0-240) for CHF6001, CHF5956 and CHF6095
Pharmacokinetic parameter (AUC0-∞) | Over 240 hours after administration in blood
  Area under plasma concentration from 0 to infinity(AUC0-∞) for CHF6001, CHF5956 and CHF6095
Pharmacokinetic parameter (tmax) | Over 240 hours after administration in blood
  Time of the maximum plasma concentration (tmax) for CHF6001, CHF5956 and CHF6095
Pharmacokinetic parameter (t1/2) | Over 240 hours after administration in blood
  Terminal half-life (t1/2) for CHF6001, CHF5956 and CHF6095
Pharmacokinetic parameter (CL/F) | Over 240 hours after administration in blood
  Apparent systemic clearance (CL/F) for CHF6001
Pharmacokinetic parameter (AUCt) | Over 240 hours after administration in blood
  Area under the plasma concentration versus time curve (AUCt) for CHF5956 and CHF6095
Pharmacokinetic parameter (Cmax) | Over 240 hours after administration in blood
  Peak Plasma Concentration (Cmax) for CHF5956 and CHF6095

CONTACTS AND LOCATIONS:
Locations (1):
- MC Comac Medical Ltd., Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piccinno A, Pittelli MG, Balzano D, Rizzo E, Bellatti P, Rostello C, Emirova A. Evaluating the Impact of Hepatic or Renal Impairment on Tanimilast (CHF6001) Pharmacokinetics: Two Open-Label, Parallel-Group, Single-Center Studies. Clin Transl Sci. 2025 May;18(5):e70261. doi: 10.1111/cts.70261. PMID 40391696